CLINICAL TRIAL: NCT04247087
Title: Effects of Fhytomenadione on Coronary Artery Calcification of Hemodialysis Patients. Randomized Clinical Trial
Brief Title: Effects of Fhytomenadione on Coronary Artery Calcification of Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Marco Antonio Ocampo Apolonio (Unknown); Rodolfo Guardado Mendoza (Unknown); Texar Alfonso Pereyra Nobara (Unknown)
Responsible Party: Principal Investigator, Hilda Elizabeth Macias Cervantes, Doctor, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Coronary Calcification
Keywords: coronary calcification; phytomenadione; chronic kidney disease; hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Vitamin K 1; Vitamin K; Solutions; Injections

STUDY DESIGN:
Intervention Model Description: randomized clinical trial with double blinding compared to placebo
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were randomly assigned to receive intravenous vitamin K or placebo solution. Coronary tomography was performed and interpreted by Radiology staff, who had no knowledge about the study groups or their intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): phytomenadione 10 mg (1 vial in the venous line of the extracorporeal hemodialysis circuit) post hemodialysis 3 times a week for 12 months
  Interventions: Drug: phytomenadione
- Control group (Placebo Comparator): 1 vial of placebo solution (solution for injection in the venous line of the extracorporeal hemodialysis circuit) post hemodialysis 3 times a week for 12 months
  Interventions: Drug: placebo solution

INTERVENTIONS:
Drug: phytomenadione — phytomenadione 10 mg (1 vial in the venous line of the extracorporeal hemodialysis circuit) post hemodialysis 3 times a week for 12 months
  Other Names: vitamin K
  Arms: Intervention group
Drug: placebo solution — 1 vial of placebo solution (solution for injection in the venous line of the extracorporeal hemodialysis circuit) post hemodialysis 3 times a week for 12 months
  Other Names: solution for injection
  Arms: Control group

SUMMARY:
Until 2013 the reported incidence of chronic kidney disease varied widely between countries, reporting the highest prevalence Taiwan, the region of Jalisco in Mexico and United States, with 458, 421 and 363 individuals per million inhabitants respectively. Mexico has around 52,000 patients in replacement therapies, of which 80% of patients are treated in the Instituto Mexicano del Seguro Social (IMSS).

In each stage of renal disease the principal cause of mortality is cardiovascular disease. The risk of cardiovascular mortality is greater than the general population. Arterial calcification, a marker of atherosclerosis and cardiovascular mortality predictor is common in chronic kidney disease. The presence of arterial calcification leads to an increase in arterial stiffness and to a decrease in coronary perfusion resulting in cardiac hypertrophy and myocardial ischemia.

The presence of traditional cardiovascular risk factors like diabetes, hypertension, hyperlipidemia and old age cannot fully explain the high prevalence of atherosclerosis and arterial calcification in chronic kidney disease. Another specific factors related to chronic kidney disease, like hyperphosphatemia, high calcium concentration in dialysis solutions, use of high doses of vitamin D for the management of hyperparathyroidism has been shown to positively influence development of arterial calcification. Invitro studies show that in presence of hyperphosphatemia smooth muscle cells are transformed into osteoblast-like cells that can express proteins that regulate mineralization. Two of this proteins, the matrix Gla protein (MGP) and osteocalcin (OC) are regulators of tissue mineralization in arterial walls and bones respectively. Vitamin K is required as cofactor in the gamma-carboxylation process of several extracellular matrix proteins, converting inactive carboxylated proteins to carboxylated active proteins. Prothrombin and coagulation factors 7,9 y 10 require vitamin K2 for its carboxylation process, while osteocalcin and the matrix Gal protein require vitamin K1. Matrix Gla protein is a calcification inhibitor that plays an important role in the prevention of arterial calcification. For carboxylation and correct function of the MGP is necessary an enzymatic cofactor, vitamin K; this is corroborated in the fact that the antagonism of vitamin K with warfarin antagonizes the carboxylation of MGP and produces rapid arterial calcification.

There are currently no studies evaluating vitamin K in the prevention of vascular calcification in patients with chronic kidney disease, therefore, the role of vitamin K in the patient with kidney disease needs to be clarified with randomized controlled studies, in which the target will be this population of patients at high risk. The aim of this study is evaluate the effect of phytomenadione on coronary artery calcification of patients on hemodialysis compared to placebo, our research hypothesis is that phytomenadione slows the progression and favors the regression of coronary arterial calcification in patients on hemodialysis compared to placebo, evaluating the coronary calcium score by coronary tomography. As secondary objectives was determine changes in the baseline coronary calcium score and at 12 months of use of phytomenadione and presence of cardiovascular events like acute myocardial infarction, unstable angina and death of cardiac cause. The intervention group received phytomenadione 10 mg (1 vial in the venous line of the extracorporeal hemodialysis circuit) post hemodialysis 3 times a week for 12 months and the control group 1 vial of placebo solution (solution for injection in the venous line of the extracorporeal hemodialysis circuit) post hemodialysis 3 times a week for 12 months. The follow-up of the patients was for 12 months, at the end of the follow-up, a coronary control tomography was performed by the Radiology Department to assess the final calcium score. Relative risk measurement (RR), absolute risk reduction (ARR) and number to be treated (NTT) were performed.

DETAILED DESCRIPTION:
In our hospital (Unidad Medica de Alta Especialidad No. 1 Bajío), there are about 130 patients on hemodialysis and estimation of cardiovascular risk is done through basic studies as the lipid profile, electrocardiogram and echocardiogram and its management is determined by classical interventions like diabetes control, hypertension and statins use, which have not shown an increase in patient survival, and it is clear that more dramatic interventions to normalize phosphate, such as intensive dialysis and even renal transplantation, cannot reverse vascular calcification. This may be because the reversion process needs to be activated at the cellular level, interventions such as the use of vitamin K as a strong tissue calcification inhibitor can be an active tool for the reversal of vascular calcification in chronic kidney disease.

By demonstrating a reversal of coronary calcification with the use of vitamin K, the incidence of cardiovascular events can be reduced, thus decreasing the progression of coronary atherosclerosis and the risk of acute myocardial infarction. The use of vitamin K may represent an economic intervention that could be implemented in the other hospital centers as a primary part of management in patients with chronic kidney disease in hemodialysis. Based on this we ask the following research question: ¿What is the effect of phytomenadione on the calcification of coronary arteries in patients on hemodialysis compared to placebo?. Our research hypothesis was that phytomenadione slows the progression and favors the regression of coronary arterial calcification in patients on hemodialysis compared to placebo.

A randomized clinical trial was designed with double blinding compared to placebo, the type of sampling was simple random probabilistic and the universe of study patients on hemodialysis of the Unidad Médica de Alta Especialidad No. 1 Bajío, with diagnosis of chronic kidney disease of any etiology that meet the tomographic criterion of a coronary calcium score of 10 Agatston units.

The selection criteria were as follows:

Inclusion criteria:

Patients with chronic kidney disease in hemodialysis Patients who have 6 months or more on hemodialysis Patients over 18 years Patients that meet the tomographic criterion of a coronary calcium score of 10 Agatston units.

Male and female right-holders of the IMSS

No Inclusion criteria:

Patients in previous or current treatment with phytomenadione Coronary stent patients Patients with arrhythmias and requiring oral anticoagulation with warfarin or acenocoumarin Pregnant patients

Exclusion criteria:

Patients who undergo renal transplantation during the follow-up period Patients who change the modality to peritoneal dialysis during the follow-up period

Elimination criteria:

Patients who wish to leave the study Patients allergic to vitamin K The start date of the study was after approval by the Electronic Registration System of the Health Research Coordination (SIRELCIS by its acronym in spanish) until the entire universe is completed and 12 months follow-up of the intervention. This work was approved by the local research and ethics committee, approved with the registration number R-2017-501-16.

The sample size was calculated based on the article by Block et al (2005) where the annual proportion of coronary artery calcification in patients on hemodialysis was evaluated with placebo use, which was 88%. Assuming that with the use of vitamin K the proportion of patients presenting with progression of coronary artery calcification will be 70%, plus an alpha error of 0.05, a test power of 80% and a single tail, a size of 27 patients per group was obtained, considering a loss of 10% the sample was increased to 30 patients per group.

The methodology was as follows: within the population of hemodialysis patients, patients who met the inclusion criteria were sought, once the participation in the study was accepted and an informed consent was signed, a coronary tomography was performed and, after completing the sample size, the patients were randomized using a random number letter.

Coronary tomography was performed and interpreted by UMAE No. 1 Radiology staff, who had no knowledge about the study groups or their intervention.

To the study group was administered 10 mg of phytomenadione (1 vial in the venous line of the extracorporeal hemodialysis circuit) post hemodialysis 3 times a week, and to the group control a placebo solution post hemodialysis 3 times a week; both vitamin K and placebo were provided by the hospital pharmacy. After each application, both the drug and the placebo were monitored for adverse effects.

The follow-up of the patients was for 12 months, at the end of the follow-up, a coronary control tomography was performed by the Radiology Department to assess the final calcium score.

The laboratory studies were processed in the hospital's laboratory and are part of the follow-up studies of patients with chronic kidney disease, they were requested upon admission of the patients in the study and at the end of the 12-month follow-up.

The results are presented with descriptive statistics with mean and standard deviation or median with confidence intervals according to the type of variable.

Qualitative variables were analyzed using Chi square or exact Fisher test. Quantitative variables using student's T or Mann Withney's W in case of not having normal distribution.

To compare coronary artery calcification between the vitamin K and placebo groups, they were compared using T from independent samples or U Mann Withney, and to compare the change between baseline and final coronary calcification in both the intervention group and the control group, the coronary calcium score delta was calculated, and a paired student's T or Wilcoxon test was performed. p values menor 0.05 were considered as significant.

Likewise, relative risk measurement (RR), absolute risk reduction (ARR) and number to be treated (NTT) were performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease in hemodialysis
* Patients who have 6 months or more on hemodialysis
* Patients over 18 years
* Patients that meet the tomographic criterion of a coronary calcium score of 10 Agatston units.

Exclusion Criteria:

* Patients in previous or current treatment with phytomenadione
* Coronary stent patients
* Patients with arrhythmias and requiring oral anticoagulation with warfarin or acenocoumarin
* Pregnant patients
* Patients who undergo renal transplantation during the follow-up period
* Patients who change the modality to peritoneal dialysis during the follow-up period
* Patients who are known allergy to vitamin K

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
coronary calcium score | 12 months
  Within the population of hemodialysis patients, patients who met the inclusion criteria were sought, once the participation in the study was accepted and an informed consent was signed, a coronary tomography was performed and interpreted by Radiology staff, who had no knowledge about the study groups or their intervention. Those patients who fulfilled the coronary calcification tomographic criterion defined as coronary calcium score of 10 Agatston units were randomized to receive the intervention or the placebo. At the end of the 12 month follow-up, a coronary tomography was performed again to quantify the final Agatston score

SECONDARY OUTCOMES:
cardiovascular events | 12 months
  determine presence of cardiovascular events like acute myocardial infarction, unstable angina and death of cardiac cause during follow-up. The presence of events will be determined according to the clinical record in the patient's file

CONTACTS AND LOCATIONS:
Overall Officials: Hilda E Macias Cervantes, Doctor, Principal Investigator — Instituto Mexicano del Seguro Social; Marco A Ocampo Apolonio, Doctor, Study Chair — Instituto Mexicano del Seguro Social; Rodolfo Guardado Mendonza, Doctor, Study Director — Universidad de Guanajuato; Texar A Pereyra Nobara, Doctor, Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital de Alta Especialidad No. 1 Bajío, Boulevard Adolfo López Mateos esquina Insurgentes S/N, colonia Los Paraísos, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Foley RN, Parfrey PS, Sarnak MJ. Clinical epidemiology of cardiovascular disease in chronic renal disease. Am J Kidney Dis. 1998 Nov;32(5 Suppl 3):S112-9. doi: 10.1053/ajkd.1998.v32.pm9820470. No abstract available.
- [Background] Block GA, Raggi P, Bellasi A, Kooienga L, Spiegel DM. Mortality effect of coronary calcification and phosphate binder choice in incident hemodialysis patients. Kidney Int. 2007 Mar;71(5):438-41. doi: 10.1038/sj.ki.5002059. Epub 2007 Jan 3. PMID 17200680
- [Background] Goodman WG, Goldin J, Kuizon BD, Yoon C, Gales B, Sider D, Wang Y, Chung J, Emerick A, Greaser L, Elashoff RM, Salusky IB. Coronary-artery calcification in young adults with end-stage renal disease who are undergoing dialysis. N Engl J Med. 2000 May 18;342(20):1478-83. doi: 10.1056/NEJM200005183422003. PMID 10816185
- [Background] Longenecker JC, Coresh J, Powe NR, Levey AS, Fink NE, Martin A, Klag MJ. Traditional cardiovascular disease risk factors in dialysis patients compared with the general population: the CHOICE Study. J Am Soc Nephrol. 2002 Jul;13(7):1918-27. doi: 10.1097/01.asn.0000019641.41496.1e. PMID 12089389
- [Background] Pilkey RM, Morton AR, Boffa MB, Noordhof C, Day AG, Su Y, Miller LM, Koschinsky ML, Booth SL. Subclinical vitamin K deficiency in hemodialysis patients. Am J Kidney Dis. 2007 Mar;49(3):432-9. doi: 10.1053/j.ajkd.2006.11.041. PMID 17336705
- [Result] Oikonomaki T, Papasotiriou M, Ntrinias T, Kalogeropoulou C, Zabakis P, Kalavrizioti D, Papadakis I, Goumenos DS, Papachristou E. The effect of vitamin K2 supplementation on vascular calcification in haemodialysis patients: a 1-year follow-up randomized trial. Int Urol Nephrol. 2019 Nov;51(11):2037-2044. doi: 10.1007/s11255-019-02275-2. Epub 2019 Sep 17. PMID 31529295
- [Result] Geleijnse JM, Vermeer C, Grobbee DE, Schurgers LJ, Knapen MH, van der Meer IM, Hofman A, Witteman JC. Dietary intake of menaquinone is associated with a reduced risk of coronary heart disease: the Rotterdam Study. J Nutr. 2004 Nov;134(11):3100-5. doi: 10.1093/jn/134.11.3100. PMID 15514282
- [Result] Kurnatowska I, Grzelak P, Masajtis-Zagajewska A, Kaczmarska M, Stefanczyk L, Vermeer C, Maresz K, Nowicki M. Effect of vitamin K2 on progression of atherosclerosis and vascular calcification in nondialyzed patients with chronic kidney disease stages 3-5. Pol Arch Med Wewn. 2015;125(9):631-40. doi: 10.20452/pamw.3041. Epub 2015 Jul 15. PMID 26176325